CLINICAL TRIAL: NCT00182572
Title: Science-Based Treatment for Opioid-Dependent Adolescents
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: St. Luke's-Roosevelt Hospital Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DA018297 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-08-12 (Estimated); Status verified 2008-08

CONDITIONS: Opioid-Dependence Among Adolescents
Keywords: heroin; opiate; addiction; adolescent; treatment
MeSH Terms: conditions — Behavior, Addictive | interventions — Buprenorphine; Naltrexone; Behavior Therapy

INTERVENTIONS:
Drug: buprenorphine
Drug: naltrexone
Procedure: behavior therapy
Procedure: voucher-based contingency management

SUMMARY:
The purpose of this study is to evaluate ways to optimize outcomes from combined behavioral-pharmacological treatment for opioid-dependent youth.

DETAILED DESCRIPTION:
Adolescents are increasingly abusing and becoming dependent on heroin and other opioids. The number of emergency room visits related to heroin among 12-17 year olds rose almost 600%, and the self-reported prevalence of heroin use among this group more than doubled in the last decade. As a result of the increased availability of high-potency, low-cost heroin, many adolescents initiate heroin use by snorting it; however, many often then progress to injection of heroin. Despite the critical need to identify efficacious treatments for this population, virtually no research has been conducted to systematically characterize or evaluate treatment interventions for adolescent heroin and opioid abusers. We recently conducted the first controlled study funded by NIDA to systematically evaluate the efficacy of several pharmacotherapies as detoxification agents along with intensive behavioral interventions in the treatment of this population. The purpose of this study is to evaluate ways to further improve on the promising outcomes from our initial study via combined behavioral-buprenorphine treatment for opioid-dependent youth. The primary aim is to examine if improved treatment outcomes can be achieved if the duration of buprenorphine detoxification is lengthened (when the rate of decrease in buprenorphine dose is slower, withdrawal symptoms may be of reduced intensity and youth are provided with a greater opportunity to learn new skills and behaviors addressing how they might best discontinue their opiate use, prevent relapse, and meet treatment goals). A secondary aim is to examine if the provision of monetary voucher-based incentives contingent on consumption of the opioid antagonist, naltrexone, reduces rates of relapse to opiate use in adolescents post-detoxification compared to when no such incentives are provided. This analysis may provide critical empirical information regarding how to best prevent relapse to opioid use among opioid-dependent youth. Another secondary aim is to identify significant predictors of treatment outcome. We will thus conduct an exploratory evaluation of demographic, baseline drug use, psychological and other history variables that may predict successful treatment outcomes. This work may help inform the refinement of treatment interventions for various sub-populations of opioid-dependent youth. Outcome measures will include opiate and other drug abstinence, retention, opiate withdrawal symptoms, HIV risk behavior, family relationships, as well as a variety of other secondary outcome measures. We plan to collect these measures at intake, during treatment and at several post-treatment follow-up timepoints. Overall, this research will contribute new empirical information that will inform the development of effective treatment interventions for the largely unstudied and rapidly expanding population of opioid-dependent youth.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of opioid dependence
* ages 13-18 years

Exclusion Criteria:

* active psychosis
* active suicidality
* major medical problems (e.g., cardiovascular disease)
* pregnancy
* require inpatient detoxification from non-opiate drugs

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2005-07

PRIMARY OUTCOMES:
opiate use

SECONDARY OUTCOMES:
treatment retention
other drug use
HIV risk behavior
opiate agonist and withdrawal effects
psychological status
family relations
motivation to change drug use
opiate craving
criminal activity

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marsch, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (1):
- Behavioral Science Research Unit, St. Luke's Hospital, New York, New York, United States

REFERENCES:
- [Derived] Marsch LA, Moore SK, Borodovsky JT, Solhkhah R, Badger GJ, Semino S, Jarrett K, Condon KD, Rossettie K, Vincent P, Hajizadeh N, Ducat E. A randomized controlled trial of buprenorphine taper duration among opioid-dependent adolescents and young adults. Addiction. 2016 Aug;111(8):1406-15. doi: 10.1111/add.13363. Epub 2016 Apr 21. PMID 26918564